CLINICAL TRIAL: NCT06729866
Title: Electrogram Guided Pulse Field Ablation for Persistent Atrial Fibrillation
Brief Title: EGM Guided PFA for PerAF
Acronym: EGM-PFA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Liu (Other)
Responsible Party: Sponsor-Investigator, Xu Liu, Dr., Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGM-PFA for PerAF
Record Dates: First submitted 2024-12-03; First posted 2024-12-11 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-12

CONDITIONS: Persistent Atrial Fibrillation
Keywords: eletrogram guided ablation; pulse field ablation; persistent atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: In persistent atrial fibrillation patients, traget electrogram was mapped firstly , pulse field ablation of pulmonary veins, posterior wall of left atrium and target electrogram was ablated, until the atrial fibrillation converted to sinus rythm or stable atrial tachycardia. The mapping and ablation procedure was repeated until AF terminated or no target electrogram was found.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Electrogram guided pulse field ablation (Experimental): In persistent atrial fibrillation patients, traget electrogram was mapped firstly , pulse field ablation of pulmonary veins, posterior wall of left atrium and target electrogram was ablated, until the atrial fibrillation converted to sinus rythm or stable atrial tachycardia. The mapping and ablation procedure was repeated until AF terminated or no target electrogram was found.
  Interventions: Procedure: electrogram guided pulse field ablation

INTERVENTIONS:
Procedure: electrogram guided pulse field ablation — In persistent atrial fibrillation patients, traget electrogram was mapped firstly , pulse field ablation of pulmonary veins, posterior wall of left atrium and target electrogram was ablated, until the atrial fibrillation converted to sinus rythm or stable atrial tachycardia. The mapping and ablation procedure was repeated until AF terminated or no target electrogram was found.

SUMMARY:
Pulse field ablation (PFA) has shown safety and efficacy in paroxysmal atrial fibrillation (AF), while the application in persistent atrial fibrillation (PerAF) is still under investigation. The investigators' previous randomized controlled trial showed favorable outcomes with electrogram (EGM) guided radiofrequency ablation in PerAF. However, EGM-guided PFA has not yet been reported.

DETAILED DESCRIPTION:
Multiple studies have confirmed that pulse field ablation (PFA) demonstrates superior safety and efficacy in pulmonary vein isolation (PVI) for paroxysmal atrial fibrillation (PAF). However, the application of PFA in persistent atrial fibrillation (PerAF) remains in the exploratory stages. The efficacy and safety of PFA across various ablation strategies require a comprehensive evaluation. Notably, electrogram (EGM) guided PFA ablation for persistent atrial fibrillation has not yet been reported in the literature.

In the investigators' previous study on radiofrequency ablation for PerAF, the investigators observed that EGM guided ablation yielded a high success rate. Furthermore, the investigators' recent research has confirmed that intraoperative termination of atrial fibrillation using EGM guided ablation is associated with favorable long-term outcomes in patients with PerAF.

The investigators aim to explore the preliminary application of EGM guided pulse field ablation (PFA) in persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented drug-resistant symptomatic persistent AF meeting all three of the following criteria:

   1. Patient is refractory or intolerant to at least one Class I/III antiarrhythmic agent
   2. ECG-documented episode of persistent AF lasting longer than 7 days
   3. Holter within 90 days of the Enrollment Date demonstrating 24 hours of continuous AF
2. Patients who are ≥ 18 years
3. Patient participation requirements:

   1. Is willing and capable of providing Informed Consent to undergo study procedures
   2. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria:

1. AF that is:

   1. Paroxysmal (longest AF episode < 7days)
   2. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
2. Left atrial anteroposterior diameter ≥ 60 mm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
3. Any of the following cardiac conditions:

   1. Clinically significant arrhythmias other than AF, AFL or AT
   2. NYHA Class IV CHF
   3. Atrial or ventricular septal defect closure
   4. Atrial myxoma
   5. History of congenital heart disease with any residual anatomic or conduction abnormality
4. Any of the following within 3 months of enrollment:

   1. Myocardial infarction
   2. Unstable angina
   3. Percutaneous coronary intervention
   4. Heart surgery (e.g. coronary artery bypass grafting, ventriculotomy, atriotomy)
   5. Heart failure hospitalization
   6. Stroke or TIA
   7. Clinically significant bleeding
   8. Pericarditis or pericardial effusion
   9. Left atrial thrombus
5. History of blood clotting or bleeding abnormalities.
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Sensitivity to contrast media not controlled by premedication
8. Women of childbearing potential who are pregnant, lactating or not using birth control
9. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to

   1. Body mass index (BMI) > 40 transplant
   2. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
   3. Renal insufficiency with an estimated creatinine clearance < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
   4. Active malignancy or history of treated cancer within 24 months of enrollment
   5. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
   6. Clinically significant infection
   7. Predicted life expectancy less than one year
10. Current or anticipated enrollment in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
freedom from any AF/AT | freedom from any AF/AT at 3 months, 6 months and 12 months respectively after the procedure; adverse events occurring within 30 days of the index or reassessment procedures.
  The feasibility primary endpoint was defined as freedom from any AF/AT episodes lasting more than 30 seconds after the blanking period without anti-arrhythmic drugs at 3 months, 6 months and 12 months respectively after the procedure.
composite of major safety events | adverse events occurring within 30 days of the index or reassessment procedures.
  The safety endpoint is a composite of major safety events including cardiac tamponade or perforation, peripheral or organ thromboembolism, stroke or transient ischemic attack (TIA), diaphragmatic paralysis, block, pericarditis, hemolysis, myocardial infarction, PV stenosis, atrioesophageal fistula, and death. The endpoint includes events occurring within 30 days of the index or reassessment procedures.

SECONDARY OUTCOMES:
AF recurrence; | freedom from any AF at 3 months, 6 months and 12 months respectively after the procedure;
  freedom from any documented AF episode lasting more than 30 seconds after the blanking period without anti-arrhythmic drug treatment at 3 months, 6 months and 12 months respectively
AT recurrence | freedom from any AT at 3 months, 6 months and 12 months respectively after the procedure;
  Secondary outcomes included: any documented AT episode lasting more than 30 seconds after the blanking period without anti-arrhythmic drug treatment at 3 months, 6 months and 12 months respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes